CLINICAL TRIAL: NCT00368953
Title: A Prospective, Randomized, Multicenter Comparison of the Drug-Eluting Stent Systems YUKON Choice and TAXUS Liberté in Patients With Diabetes Mellitus
Brief Title: YUKON Choice Versus TAXUS Liberté in Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: Translumina GmbH (Industry)
Responsible Party: Holger Thiele, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Lipsia-Yukon-DM
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Yukon Choice stent system
- 2 (Active Comparator)
  Interventions: Device: Taxus Liberté stent system

INTERVENTIONS:
Device: Yukon Choice stent system — coronary stent implantation
  Arms: 1
Device: Taxus Liberté stent system — coronary stent implantation
  Arms: 2

SUMMARY:
Revascularisation procedures such as percutaneous coronary intervention are associated with overall worse outcomes in patients with diabetes mellitus. Implantation of coronary stents is associated with higher restenosis rates compared to non-diabetic individuals.

There is only limited data available on the efficacy and safety of the novel Yukon Choice drug-eluting stent system specifically in patients with diabetes mellitus. The trial will determine the efficacy and safety of the novel Yukon Choice stent system compared to the well established Taxus Liberté stent system. The primary endpoint will be "in-stent late lumen loss" at 9 months as determined by invasive angiography.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* diabetes mellitus
* symptoms (stable or unstable angina pectoris) or objective evidence of myocardial ischemia
* one or more de novo lesions in 1, 2 or 3 native coronary arteries
* clinically significant diameter of stenosis (50-99 % according to visual assessment of operator)
* lesion must be covered by stent length of no more than 24 mm and stent diameter of no more than 3,5 mm
* vessel diameter of no more than 4 mm in vessel area adjacent to stenosis
* informed consent

Exclusion Criteria:

* unprotected left main disease
* complete occlusion of target vessel
* in-stent-restenosis
* stenoses of bypass grafts
* indication for bypass surgery
* bifurcation lesions (side branch > 2,0 mm)
* thrombus in target lesion as visualized by angiography
* allergy or contraindication to concomitant medication (clopidogrel, aspirin, heparin, contrast media)
* acute myocardial infarction within preceding 48h
* participation in another trial
* pregnancy
* severe disorder of coagulation or platelet function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
"In-stent late lumen loss" at follow-up-angiography (9 months) | 9 months

SECONDARY OUTCOMES:
Binary restenosis | 9 months
Target vessel revascularisation rate | 9 months
Target lesion revascularisation rate | 9 months
Late loss (in-segment) | 9 months
MLD und diameter of stenosis (%) | 9 months
Death | 9 months
Success rate index procedure (residual diameter stenosis < 30%) | 0 months
Combined MACE (cardiac death, myocardial infarction, emergency bypass, stent thrombosis, target lesion revascularization) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] Stiermaier T, Heinz A, Schloma D, Kleinertz K, Danschel W, Erbs S, Linke A, Boudriot E, Lauer B, Schuler G, Thiele H, Desch S. Five-year clinical follow-up of a randomized comparison of a polymer-free sirolimus-eluting stent versus a polymer-based paclitaxel-eluting stent in patients with diabetes mellitus (LIPSIA Yukon trial). Catheter Cardiovasc Interv. 2014 Feb 15;83(3):418-24. doi: 10.1002/ccd.25131. Epub 2013 Aug 9. PMID 23873579
- [Derived] Desch S, Schloma D, Mobius-Winkler S, Erbs S, Gielen S, Linke A, Yu J, Lauer B, Kleinertz K, Danschel W, Schuler G, Thiele H. Randomized comparison of a polymer-free sirolimus-eluting stent versus a polymer-based paclitaxel-eluting stent in patients with diabetes mellitus: the LIPSIA Yukon trial. JACC Cardiovasc Interv. 2011 Apr;4(4):452-9. doi: 10.1016/j.jcin.2010.11.016. PMID 21511226